CLINICAL TRIAL: NCT05972070
Title: Integration of Telemedicine and Home-Based Cardiac Rehabilitation: Feasibility, Efficacy, and Adherence
Status: Recruiting | Type: Observational
Sponsor: ROM Technologies, INC (Industry)
Responsible Party: Sponsor
Other Study IDs: ROMTherapy_HBCR_1001
Record Dates: First submitted 2023-07-03; First posted 2023-08-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction; Percutaneous Transluminal Coronary Angioplasty; Coronary Artery Bypass; Stable Angina; Heart Failure; Valve Disease, Heart; Cardiac Rehabilitation; Stent
Keywords: Cardiac rehabilitation; Home based cardiac rehabilitation; Telemedicine and Home-Based Cardiac Rehabilitation
MeSH Terms: conditions — Myocardial Infarction; Angina, Stable; Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Cardiac patients: Adult patients who have undergone surgical or percutaneous coronary revascularization due to atherosclerotic coronary artery disease.
  Interventions: Device: ROMTech Portable Connect

INTERVENTIONS:
Device: ROMTech Portable Connect — The ROMTech PortableConnect Rehab System is a continuous rehabilitative exercise therapy device that uses assisted movement to measure, evaluate, exercise, re-educate and strengthen muscles, and to increase joint range of motion.
  Other Names: ROMTech PC; ROMTech PortableConnect Rehab System

SUMMARY:
The aim of this study is to evaluate feasibility, efficacy, and adherence of home-based cardiac rehabilitation with the integration of telemedicine. Several components will be assessed such as quality-of-life, nutritional counseling, maximum metabolic activity (MET's), diabetic management, tobacco cessation, lipid, blood pressure, and psychosocial management. These tasks will be accomplished through concurrent conversations between patients and their therapist's utilizing telemedicine with observed exercise training.

DETAILED DESCRIPTION:
The focus of this study is to determine the feasibility, efficacy, and adherence of home-based cardiac rehabilitation with the integration of telemedicine. The study consists of an initial review, rehabilitation sessions, nutrition consultation, and risk stratification. Once the patient is cleared for the rehabilitation program, they will be assigned a cardiac rehab specialist and begin the 36 rehabilitation sessions. The sessions include pre-session questions, surveys, pre-, during, and post vitals, exercise protocol, and off-the-device exercises.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18
2. NYHA Functional Class I, II,
3. Recent (within 60 days) status post coronary artery revascularization for atherosclerotic coronary artery disease (coronary artery bypass grafting or percutaneous coronary revascularization with stent implantation)
4. Candidate for traditional center-based cardiac rehabilitation

Exclusion Criteria:

1. Under the age of 18
2. Adults lacking capacity to consent.
3. NYHA Functional Class III, IV
4. Acute coronary syndrome
5. Systolic heart failure (LV EF <40%)
6. Status post cardiac surgery for structural heart disease or heart transplant
7. Percutaneous coronary angioplasty
8. Adults lacking capacity to consent.
9. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have undergone surgical or percutaneous coronary revascularization due to atherosclerotic coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Session attended | 12 weeks (End of treatment)
  Measure the number of sessions attended to determine the ease of patients to utilize home-based cardiac rehab integrated with telemedicine (non-inferiority to historical controls)
Sessions completed | 12 weeks(End of treatment)
  Measure the number of sessions completed to determine compliance of patients to utilize home-based cardiac rehab integrated with telemedicine
Duke Activity Status Index (DASI) | Baseline, 12 weeks (End of Treatment)
  Estimate of functional capacity
Patient Health Questionnaire(PHQ) | Baseline, 12 weeks (End of Treatment)
  Quality of Life assessment
Short Physical Performance Battery | Baseline, 12 weeks (End of Treatment)
  Lower extremity functional assessment
Short Form-36 | Baseline, 12 weeks (End of Treatment)
  Quality of Life assessment

SECONDARY OUTCOMES:
Laboratory assessment | Baseline, 12 weeks (End of Treatment)
  To determine if there is an improvement in low density lipoprotein, triglycerides,

CONTACTS AND LOCATIONS:
Locations (1):
- ROMTech, Brookfield, Connecticut, United States